CLINICAL TRIAL: NCT03945578
Title: Effects of Visceral Manipulation Associated With Pelvic Floor Muscles Training in Women With Urinary Incontinence: a Randomized Controlled Trial
Brief Title: Effects of Visceral Manipulation in Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Clinical Professor, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Visceral Manipulation
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): This group performed a supervised Pelvic Floor Muscle Training (PFMT) protocol associated with a manual sham therapy (MST) sessions.
  The PFMT protocol consisted of 20 sessions of 45-60 minutes each, twice a week, totalizing a five weeks treatment.
  The MST protocol was performed once a week, during five weeks lasting approximately 15 minutes.
  Interventions: Other: Pelvic Floor muscle training - PFMT; Other: Manual Sham Therapy - MST
- Experimental Group (Experimental): The experimental group performed the same PFMT protocol as the CG, but associated with a Visceral Manual Therapy (VMT) protocol.
  The VMT sessions were held once a week, for five weeks. Each session lasted approximately 20 minutes.
  Interventions: Other: Pelvic Floor muscle training - PFMT; Other: Visceral Manual Therapy - VMT

INTERVENTIONS:
Other: Pelvic Floor muscle training - PFMT — Pelvic Floor muscle training is an active exercise-based treatment designed to strengthen the pelvic floor muscles. The PFMT protocol was divided into four phases. Proprioceptive (2 weeks): where the woman has gained adequate perception of PFM and control of fast and slow contractions; Simple (1 week): performed with the objective of promoting control of fast and slow contractions associated with small functional exercises; Elaborated (1 week): where the exercise evolved into functional exercises of greater amplitude; and Power (1 week): where the control of the pelvic floor was promoted during efforts. In all sessions, contractions were performed for slow and for fast fibers (the list of exercises and a detailed description of them is in Appendix 1).
Other: Visceral Manual Therapy - VMT — Visceral manual therapy:is a manual treatment intended to the release of visceral fascias. The VMT protocol was based on the work proposed by Vanderheyden-Busquet (2014). To act on the abdominal and pelvic visceral fasciae, the VMT was performed through slow and deep mobilizations, respecting the participant's tissue resistance and painful response, in different regions of the abdômen.
  Arms: Experimental Group
Other: Manual Sham Therapy - MST — The manual sham therapy protocol was perfomed by gentle techniques applied to the thoracic spine, scapular waist and cervical spine
  Arms: Control Group

SUMMARY:
The objective of the study is to compare the effects of visceral manual therapy associated with pelvic floor muscle training on urinary incontinence symptoms, vaginal resting pressure and maximum voluntary contraction of the pelvic floor muscles in women. This is a randomized controlled trial with double blinding. Participants will be randomized into two groups: control and experimental. Both groups will undergo a pelvic floor muscle training program twice weekly for 5 consecutive weeks. Participants in the intervention group will also receive, once a week, a visceral manual therapy protocol and control group participants will receive a manual sham therapy protocol.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled trial with two groups. Participants will be evaluated by a trained blinded investigator and assigned randomly to the experimental and control groups. Both groups will undergo a pelvic floor muscle training program twice weekly for 5 consecutive weeks. Participants in the intervention group will also receive, once a week, a visceral manual therapy protocol and control group participants will receive a sham manual therapy protocol. Participants who agree to participate in the survey will sign a Free and Informed Consent Form and will be informed of the possibility of withdrawing from the survey at any stage, without penalty. The collection of the evaluation and intervention will be carried out in a salon Clinic School of Physiotherapy in the Center of Health and Sports Sciences (CEFID) of the State University of Santa Catarina (UDESC) in the city of Florianópolis - SC. All personal identification data of the participants will be preserved according to resolution of the national health council, taking into account the possibility of scientific dissemination of the results obtained. The risks of these procedures will be medium, since the participant may present muscle pain after the intervention protocol. To minimize these risks will be available, if necessary, attendance at the Clinic School of Physiotherapy. The sample will be selected in a non-probabilistic way for convenience. The participants will Female volunteers , aged from 18 years with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria: having a pre-established complaint or diagnosis of UI symptoms (assessed using the International Consultation on Incontinence Questionnaire - Short Form - ICIQ-UI-SF), age ≥ 18 years, have not undergone drug treatment for UI for at least 6 months; and have not previously performed surgical procedure for UI or PFMT in the 6 months before the research.

Exclusion Criteria: diagnosis or signs and symptoms of neurological diseases (self-report), BMI ≥35, gestational period, ongoing gynecological disease, initiate drug treatment for UI during the research, not reaching 80% attendance at intervention sessions, pelvic organs prolapse with a degree greater than II, absence of pelvic floor muscle contraction during assessment, known aortic aneurysm, acute inflammatory phase of gastrointestinal or genitourinary tract diseases, any other contraindication to performed VMT, or any other condition that would limit the execution of VMT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptoms of urinary incontinence and its impact on quality of life | Pre intervention, week 3 and 1 week post intervention
  This outcome will be measured through the International Consultation on Incontinence Questionnaire - Short Form. This is a self-administered questionnaire designed to assess the frequency, severity, and impact of urinary incontinence on the quality of life of patients of both sexes. It consists of four items. The first three assess the frequency, severity, and impact of urinary incontinence on quality of life. From the sum of these three items the total score is obtained, which can vary between 0 and 21 points. The higher the score, greater the severity of the symptoms of urinary incontinence. The overall score can be divided into four severity categories: mild (1-5 points), moderate (6-12 points), severe (13-18 points), very severe (19-21 points). The fourth item does not enter the total score but serves to determine the type of urinary incontinence (stress, urgency or mixed).

SECONDARY OUTCOMES:
Change from baseline in vaginal resting pressure | Pre intervention and 1 week post intervention
  this outcome will be measured by digital perineometer - Peritron 9300®
Change from baseline in maximum voluntary contraction of the pelvic floor muscles | Pre intervention and 1 week post intervention
  this outcome will be measured by digital perineometer - Peritron 9300®

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health and Sport Sciences of the State University of Santa Catarina, Florianópolis, Santa Catarina, Brazil